CLINICAL TRIAL: NCT05089604
Title: Tacrolimus Associated Tremors in Liver Transplant Recipients: a Randomized Open Label Trial Comparing De Novo Extended-release Once Daily (LCP-TAC) and Twice Daily Immediate-release (IR-TAC) Tacrolimus Formulations
Brief Title: Tacrolimus Associated Tremors in Liver Transplantation: Immediate-Release Versus Extended-Release Formulations
Acronym: LCP-TAC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Paladin Labs Inc. (Other)
Responsible Party: Principal Investigator, Trana Hussaini, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-01688
Record Dates: First submitted 2021-10-08; First posted 2021-10-22 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Liver Transplantation; Immunosuppression; Neurotoxicity; Tremor; Tacrolimus
Keywords: Liver Transplant; Tacrolimus; Immunosuppression; Tremor; Envarsus; LCP-TAC; Neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes; Tremor | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCPT (Experimental)
  Interventions: Drug: Tacrolimus Extended Release Oral Tablet
- IR-TAC (Active Comparator)
  Interventions: Drug: Tacrolimus, Immediate Release, Oral

INTERVENTIONS:
Drug: Tacrolimus, Immediate Release, Oral — Twice Daily Tacrolimus
  Other Names: Tacrolimus, Sandoz; Prograf
  Arms: IR-TAC
Drug: Tacrolimus Extended Release Oral Tablet — Once Daily Tacrolimus
  Other Names: Envarsus
  Arms: LCPT

SUMMARY:
This is a randomized open label study in de novo liver transplant recipients that aims to compare the risk of tacrolimus induced tremors with once daily extended-release formulation, Envarsus, versus the twice daily immediate-release formulation. Both formulations of tacrolimus are currently approved for the prevention of rejection in liver transplant patients.

DETAILED DESCRIPTION:
Purpose: This study is designed to evaluate the incidence and severity of tremors with two different tacrolimus formulations (LCPT versus IR-TAC) when administered in combination with mycophenolate and short term corticosteroids in de novo liver transplant (LT) recipients.

Hypothesis: In de novo liver transplant recipients, an LCPT-based immunosuppression regimen, in combination with mycophenolate and short term steroids offers improved neurotoxicity profile as evidenced by lower incidence and severity of tremors and treatment discontinuation when compared to an identical regimen using twice-daily immediate-release tacrolimus.

Rationale: Tacrolimus is the first line immunosuppressive agent in all organ transplantation and its use is associated with improved patient and graft outcomes. Neurotoxicity including headaches and tremors are amongst common dose limiting toxicities associated with tacrolimus early after liver transplantation. Mitigation strategies include dosage reduction or switch to CSA, both of which can put patient at risk of rejection and other toxicities. LCPT is a new extended release formulation with improved PK parameters and evidence of improved tolerability (lower risk of tremors) in renal transplant population. In this study, we will compare the incidence and severity of tremors associated with IR-TAC, which is currently standard of care at our institution, with LCPT, which is a new dosage form added to the hospital formulary. We will be using wearable sensors to assess the severity of tremors. Furthermore, the objective and systematic documentation of tremor severity during the first 8 weeks after transplantation will provide granular data that will elucidate the natural history of tacrolimus induced tremors early post liver transplantation.

Research design: This is a single centre, prospective, randomized, open label, parallel group trial in adult de novo liver transplant recipients. Patients will be randomized (1:1) to either LCPT or IR-TAC, both groups will receive mycophenolate and short term steroids according to the standard of care protocol. This is a superiority study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older
2. Recipients of a first-time liver transplant
3. eGFR more than 30 ml/min on the day of tacrolimus initiation
4. All patients who are eligible to initiate Tacrolimus within 7 days post-liver transplant
5. Informed consent

Exclusion Criteria:

1. Recipients of prior organ transplant
2. Need for hemodialysis either prior or following liver transplantation
3. Recipients of living donor liver or split deceased donor liver allografts
4. Recipients of combined liver/kidney transplants
5. Recipients receiving liver allografts from donors with HCV viremia (detected through nucleic acid testing or other means)
6. Patients with a history of tremor prior to transplantation including essential tremors, Parkinson's or Parkinsonian syndromes
7. Patients receiving concomitant medications known to induce tremors such as dopamine blocking agents
8. Baseline TSH, T3, T4 indicating hyperthyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with tacrolimus induced tremors or worsening tremors or tacrolimus discontinuation due to neurotoxicity at 8 weeks post transplantation | 8 weeks post transplantation
  Composite end point of proportion of patients with new tremor as defined by Kinesia One average score of 1 or greater or an increase from baseline of greater than or equal to 1 point at week 8 after transplantation, or tacrolimus discontinuation due to neurotoxicity (tremor, headaches, seizure or dysarthria).

SECONDARY OUTCOMES:
Proportion of patients reaching the composite end point of death, graft loss or biopsy proven acute cellular rejection (BPAR) at 12 months post transplantation | 12 months post transplantation
  The proportion of patients reaching the composite end point of death, graft loss or biopsy proven acute cellular rejection (BPAR)
Tremor related quality of life satisfaction as assessed by the Quality of Life in Essential Tremor (QUEST) scale | 8 weeks post transplantation
  The Quality of Life in Essential Tremor (QUEST) is a 30 item scale rated on five-point scale (0-4), corresponding to the frequency (never, rarely, sometimes, frequently, always) with scores ranging from 0 to 120. Higher scores indicate greater dissatisfaction or disability.
Immunosuppression medication adherence as assessed by the Simplified Medication Adherence Questionnaire (SMAQ) at 8 weeks after transplant | 8 weeks post transplant
  Simplified Medication Adherence Questionnaire (SMAQ) consists of six questions evaluating different aspects of patient adherence, such as forgetfulness, routine and adverse events. SMAQ is a self-reported questionnaire that has been validated in transplant population. Patients are considered adherent if they reply to all questions with an adherent answer in all six SMAQ items. (ie 1-"yes" , 2-4 - "no", not having missed more than 2 doses during last week or having failed to take the medication on not more than 2 days during the last 3 months.
  We are measuring SMAQ twice for this study (at 8 weeks and again at 12 months). Based on the literature, transplant patients are more likely to be adherent early after transplantation but they become progressively less adherent with time after transplant. We would like to determine if once daily tacrolimus has any impact on adherence.
Immunosuppression medication adherence as assessed by the Simplified Medication Adherence Questionnaire (SMAQ) at 12 months after transplant | 12 months post transplantation
  Simplified Medication Adherence Questionnaire (SMAQ) consists of six questions evaluating different aspects of patient adherence, such as forgetfulness, routine and adverse events. SMAQ is a self-reported questionnaire that has been validated in transplant population. Patients are considered adherent if they reply to all questions with an adherent answer in all six SMAQ items. (ie 1-"yes" , 2-4 - "no", not having missed more than 2 doses during last week or having failed to take the medication on not more than 2 days during the last 3 months.
  We are measuring SMAQ twice for this study (at 8 weeks and again at 12 months). Based on the literature, transplant patients are more likely to be adherent early after transplantation but they become progressively less adherent with time after transplant. We would like to determine if once daily tacrolimus has any impact on adherence.

OTHER OUTCOMES:
Incidence of biopsy proven acute cellular rejection (BPAR) | 3, 6 and 12 months post transplantation
  Incidence of biopsy proven acute cellular rejection (BPAR) by Banff 97 criteria
Incidence and severity of AKI | 1,3 and 6 months post transplant
  Incidence and severity of AKI based on KDIGO classification
eGFR (MDRD) < 45 mL/min and < 30 mL/min | 6 & 12 months after transplant
  Proportion of patients with eGFR (MDRD) < 45 mL/min and < 30 mL/min
Change in GFR | 12 months after transplant
  Change in GFR from month 1 (day 28) to month 12 (day 364)
Incidence of new onset diabetes after transplantation (NODAT) | 6 and 12 months post transplant
  Incidence of new onset diabetes after transplantation (NODAT)
Severity of tremors | 2, 4, 6 and 8 weeks after transplantation
  Proportion of patients with mild, moderate and severe tremor

CONTACTS AND LOCATIONS:
Overall Officials: Trana Hussaini, Pharm D, Principal Investigator — University of British Columbia; Jo-Ann Ford, RN, Study Chair — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided